CLINICAL TRIAL: NCT02089217
Title: Carotid Revascularization and Medical Management for Asymptomatic Carotid Stenosis Trial
Acronym: CREST-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, James F. Meschia, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 13-004051; U01NS080168 (NIH)
Record Dates: First submitted 2014-03-13; First posted 2014-03-17 (Estimated); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Carotid Stenosis
Keywords: asymptomatic; carotid; stent; endarterectomy; embolic protection; medical management; hypertension; hyperlipidemia; cognition; risk factor control
MeSH Terms: conditions — Carotid Stenosis; Hypertension; Hyperlipidemias | interventions — Endarterectomy, Carotid

STUDY DESIGN:
Intervention Model Description: CREST-2 is two parallel multi-center randomized, observer-blinded endpoint clinical trials.
Who Masked: Investigator
Masking Description: CREST-2 is two parallel multi-center randomized, observer-blinded endpoint clinical trials.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Carotid Endarterectomy (CEA) (Active Comparator): Carotid Endarterectomy
  Interventions: Procedure: Carotid endarterectomy (CEA)
- Carotid Stenting (CAS) (Active Comparator): Carotid Stenting
  Interventions: Device: Carotid Stenting (CAS)
- Intensive Medical Management - no CEA (Experimental): Intensive Medical Management alone - no CEA
  Interventions: Other: Intensive Medical Management - no CEA
- Intensive Medical Management - no CAS (Experimental): Intensive Medical Management alone - no CAS
  Interventions: Other: Intensive Medical Management - no CAS

INTERVENTIONS:
Procedure: Carotid endarterectomy (CEA) — Carotid endarterectomy
  Arms: Carotid Endarterectomy (CEA)
Device: Carotid Stenting (CAS) — Carotid stenting
  Arms: Carotid Stenting (CAS)
Other: Intensive Medical Management - no CEA — Intensive Medical Management alone - no CEA
  Arms: Intensive Medical Management - no CEA
Other: Intensive Medical Management - no CAS — Intensive Medical Management alone - no CAS
  Arms: Intensive Medical Management - no CAS

SUMMARY:
Carotid revascularization for primary prevention of stroke (CREST-2) is two independent multicenter, randomized controlled trials of carotid revascularization and intensive medical management versus medical management alone in patients with asymptomatic high-grade carotid stenosis. One trial will randomize patients in a 1:1 ratio to endarterectomy versus no endarterectomy and another will randomize patients in a 1:1 ratio to carotid stenting with embolic protection versus no stenting. Medical management will be uniform for all randomized treatment groups and will be centrally directed.

DETAILED DESCRIPTION:
Prevention of stroke involves managing and treating risk factors. Most strokes are caused when blood flow to a portion of the brain is blocked. One place this often happens is in the carotid artery. This blockage is called atherosclerosis or hardening of the arteries.

The purpose of this trial is to determine the best way to prevent strokes in people who have a high amount of blockage of their carotid artery but no stroke symptoms related to that blockage. Each eligible participant will be evaluated to determine which procedure(s) is best for him/her. All participants will receive intensive medical treatment. In addition, participants will be randomized to receive the selected procedure or not.

The trial will be conducted in the United States and Canada by physicians carefully selected on their ability to perform the procedures at low risk. Another key component of the trial is that important stroke risk factors, including hypertension, diabetes, high cholesterol, cigarette smoking, physical activity, and diet will be managed intensively. Participants will remain in the study for 4 years.

ELIGIBILITY:
General Inclusion Criteria

1. Patients ≥35 years old.
2. Carotid stenosis defined as:

   * Stenosis ≥70% by catheter angiography (NASCET Criteria); OR
   * by Doppler ultrasonography (DUS) with ≥70% stenosis defined by a peak systolic velocity of at least 230 cm/s plus at least one of the following:

     1. an end diastolic velocity ≥100 cm/s, or
     2. internal carotid/common carotid artery peak systolic velocity ratio ≥4.0, or
     3. computed tomography angiography (CTA) with ≥ 70% stenosis, or
     4. magnetic resonance angiography (MRA) with ≥ 70% stenosis.
3. No medical history of stroke or transient ischemic attack (TIA) ipsilateral to the stenosis within 180 days of randomization. Life-long asymptomatic patients will be defined as having no medical history of stroke or transient ischemic attack and negative responses to all of the symptom items on the Questionnaire for Verifying Stroke-free Status (QVSS).
4. Patients must have a modified Rankin Scale (mRS) score of 0 or 1 at the time of informed consent.
5. Women must not be of childbearing potential or, if of childbearing potential, have a negative pregnancy test prior to randomization.
6. Patients must agree to comply with all protocol-specified follow-up appointments.
7. Patients must sign a consent form that has been approved by the local governing Institutional Review Board (IRB)/Medical Ethics Committee (MEC) of the respective clinical site.
8. Randomization to treatment group will apply to only one carotid artery for patients with bilateral carotid stenosis. Management of the non-randomized stenosis may be done in accordance with local PI recommendation. Treatment of the non-study internal carotid artery must take place at least 30 days prior to randomization, or greater than 44 days after randomization and 30 days after the study procedure is completed (whichever is longer).
9. Carotid stenosis must be treatable with carotid endarterectomy (CEA), carotid artery stenting (CAS), or either procedure.

General Exclusion Criteria

1. Intolerance or allergic reaction to a study medication without a suitable management alternative.
2. GI hemorrhage within 1 month prior to enrollment that would preclude antiplatelet therapy.
3. Prior major ipsilateral stroke in the past with substantial residual disability (mRS ≥ 2) that is likely to confound study outcomes.
4. Severe dementia.
5. History of major symptomatic intracranial hemorrhage within 12 months that was not related to anticoagulation.
6. Prior Intracranial hemorrhage that the investigator believes represents a contraindication to the perioperative or periprocedural antithrombotic and antiplatelet treatments necessary to complete endarterectomy or stenting per protocol.
7. Current neurologic illness characterized by fleeting or fixed neurologic deficits that cannot be distinguished from TIA or stroke.
8. Patient objects to future blood transfusions.
9. Platelet count <100,000/microliter or history of heparin-induced thrombocytopenia.
10. Anticoagulation with Phenprocoumon (Marcumar®), warfarin, or a direct thrombin inhibitor, or anti-Xa agents.
11. Chronic atrial fibrillation, unless the patient has had successful atrial appendage closure (e.g., Watchman Device) and no longer requires chronic therapeutic anticoagulation.
12. Any episode of atrial fibrillation within the past 6 months or history of paroxysmal atrial fibrillation that is deemed to require chronic anticoagulation.
13. Other high-risk cardiac sources of emboli, including left ventricular aneurysm, severe cardiomyopathy, aortic or mitral mechanical heart valve, severe calcific aortic stenosis (valve area < 1.0 cm2), endocarditis, moderate to severe mitral stenosis, left atrial thrombus, or any intracardiac mass, or known unrepaired patent foramen ovale (PFO) with prior paradoxical embolism.
14. Unstable angina defined as rest angina with electrocardiogram (ECG) changes that is not amenable to revascularization (patients should undergo planned coronary revascularization at least 30 days before randomization).
15. Left Ventricular Ejection fraction <30% or admission for heart failure in prior 6 months.
16. Respiratory insufficiency with life expectancy < 4 years or forced expiratory volume (FEV1) <30% of predicted value.
17. Known malignancy other than basal cell non-melanoma skin cancer. There are two exceptions to this rule: patients with prior cancer treatment and no recurrence for >5 years are eligible for enrollment and cancer patients with life expectancy of greater than 5 years are eligible for enrollment.
18. Any major surgery, major trauma, revascularization procedure, or acute coronary syndrome within the past 1 month.
19. Either the serum creatinine is ≥ 2.5 mg/dl or the estimated glomerular filtration rate (GFR) is < 30 cc/min.
20. Major (non-carotid) surgery/procedures planned within 3 months after enrollment.
21. Currently listed or being evaluated for major organ transplantation (i.e. heart, lung, liver, kidney).
22. Actively participating in another drug or aortic arch or cerebrovascular device trial for which participation in CREST-2 would be compromised with regard to follow-up assessment of outcomes or continuation in CREST-2.
23. Inability to understand and cooperate with study procedures or provide informed consent.
24. Non-atherosclerotic carotid stenosis (dissection, fibromuscular dysplasia, or stenosis following radiation therapy).
25. Previous ipsilateral CEA or CAS.
26. Ipsilateral internal or common carotid artery occlusion.
27. Intra-carotid floating thrombus.
28. Ipsilateral intracranial aneurysm > 5 mm.
29. Extreme morbid obesity that would compromise patient safety during the procedure or would compromise patient safety during the periprocedural period.
30. Coronary artery disease with two or more proximal or major diseased coronary arteries with 70% stenosis that have not, or cannot, be revascularized.

Specific Carotid Endarterectomy Exclusion Criteria

Patients who are being considered for revascularization by CEA must not have any of the following criteria:

1. Serious adverse reaction to anesthesia not able to be overcome by pre-medication.
2. Distal/intracranial stenosis greater than index lesion.
3. Any of the following anatomical: radical neck dissection; surgically inaccessible lesions (e.g. above cervical spine level 2 (C2)); adverse neck anatomy that limits surgical exposure (e.g. spinal immobility - inability to flex neck beyond neutral or kyphotic deformity, or short obese neck); presence of tracheostomy stoma; laryngeal nerve palsy contralateral to target vessel; or previous extracranial-intracranial or subclavian bypass procedure ipsilateral to the target vessel.

Specific Carotid Artery Stenting Exclusion Criteria

Patients who are being considered for revascularization by CAS must not have any of the following criteria:

1. Allergy to intravascular contrast dye not amenable to pre-medication.
2. Type III, aortic arch anatomy.
3. Angulation or tortuosity (≥ 90 degree) of the innominate and common carotid artery that precludes safe, expeditious sheath placement or that will transmit a severe loop to the internal carotid after sheath placement.
4. Severe angulation or tortuosity of the internal carotid artery (including calyceal origin from the carotid bifurcation) that precludes safe deployment of embolic protection device or stent. Severe tortuosity is defined as 2 or more ≥ 90 degree angles within 4 cm of the target stenosis.
5. Proximal/ostial common carotid artery (CCA), innominate stenosis or distal/intracranial stenosis greater than index lesion.

   Excessive circumferential calcification of the stenotic lesion defined as >3mm thickness of calcification seen in orthogonal views on fluoroscopy.(Note: Anatomic considerations such as tortuosity, arch anatomy, and calcification must be evaluated even more carefully in elderly subjects (≥ 70 years).)
6. Target ICA vessel reference diameter <4.0 mm or >9.0 mm. Target internal carotid artery (ICA) measurements may be made from angiography of the contralateral artery. The reference diameter must be appropriate for the devices to be used.
7. Inability to deploy or utilize an FDA-approved Embolic Protection Device (EPD).
8. Non-contiguous lesions and long lesions (>3 cm).
9. Qualitative characteristics of stenosis and stenosis-length of the carotid bifurcation (common carotid) and/or ipsilateral external carotid artery, that preclude safe sheath placement.
10. Occlusive or critical ilio-femoral disease including severe tortuosity or stenosis that necessitates additional endovascular procedures to facilitate access to the aortic arch or that prevents safe and expeditious femoral access to the aortic arch. "String sign" of the ipsilateral common or internal carotid artery.
11. Angiographic, computed tomography (CT), magnetic resonance (MR) or ultrasound evidence of severe atherosclerosis of the aortic arch or origin of the innominate or common carotid arteries that would preclude safe passage of the sheath and other endovascular devices to the target artery as needed for carotid stenting.

Ages: 35 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2486 (Actual)
Dates: Start 2014-12-09 (Actual); Primary Completion 2025-09-12 (Actual); Study Completion 2025-09-12 (Actual)

PRIMARY OUTCOMES:
Stroke and death | 4 years
  The primary outcome is the composite of stroke plus death within 44 days after randomization and ipsilateral stroke thereafter up to 4 years.

SECONDARY OUTCOMES:
Cognitive Function | 4 years
  The assess if MEDICAL management differs from CAS, and differs from CEA, to maintain the level of cognitive function at the 4-year assessment.
Major Stroke | 4 years
  if there are treatment differences in the incidence of major stroke at 4-years among all arms of the study
Effect modification | 4 years
  Potential effect modification of the CAS or CEA versus MEDICAL differences, based on patient age, sex, severity of carotid stenosis, restenosis, risk factor level, and duration of asymptomatic period.

CONTACTS AND LOCATIONS:
Overall Officials: James F. Meschia, MD, Principal Investigator — Mayo Clinic; Brajesh K. Lal, MD, Principal Investigator — University of Maryland; George Howard, DrPH, Principal Investigator — University of Alabama at Birmingham; Lloyd Edwards, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (167):
- United States (154):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Huntsville Hospital/ Heart Center Research Alabama, Huntsville, Alabama
  - Banner University Medical Center, Phoenix, Arizona
  - St. Joseph's Hospital and Medical Center/Barrow Neurological Institute, Phoenix, Arizona
  - Abrazo Arizona Heart Hospital, Phoenix, Arizona
  - Mayo Clinic Arizona, Phoenix, Arizona
  - HonorHealth Scottsdale Osborn Medical Center, Scottsdale, Arizona
  - Banner University Medical Center, Tucson, Arizona
  - Central Arkansas Veteran's Healthcare System, Little Rock, Arkansas
  - Mission Cardiovascular Research Institute, Fremont, California
  - Mission Cardiovascular Research, Fremont, California
  - University of California Irvine, Irvine, California
  - UC San Diego Health, La Jolla, California
  - Kaiser Permanente Los Angeles, Los Angeles, California
  - Keck Medical Center of University of Southern California, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California Los Angeles (UCLA), Los Angeles, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - University of California San Diego, San Diego, California
  - Kaiser Permanente, San Diego, California
  - Kaiser Permanente Northern California, San Francisco, California
  - University of California San Francisco, San Francisco, California
  - San Francisco VA Medical Center, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - St. Joseph's Medical Center, Stockton, California
  - Providence Little Company of Mary Medical Center, Torrance, California
  - St. Mary's Hospital Regional Medical Center, Grand Junction, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut
  - Medstar/Washington Hospital Center, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - University of Florida Health at Shands, Gainesville, Florida
  - Lyerly Neurosurgery, Jacksonville, Florida
  - UF Jacksonville, Jacksonville, Florida
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - University of Miami Hospital, Miami, Florida
  - Miami Cardiac and Vascular Institute at Baptist Hospital of Miami, Miami, Florida
  - Mount Sinai Medical Center of Florida, Miami Beach, Florida
  - Cardiovascular Institute of Northwest Florida, Panama City, Florida
  - Tallahassee Neurological Clinic, Tallahassee, Florida
  - Tampa General/University of South Florida, Tampa, Florida
  - Atlanta VA Medical Center, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Southern Illinois Healthcare, Carbondale, Illinois
  - The University of Chicago Medical Center, Chicago, Illinois
  - Northshore University, Evanston, Illinois
  - Northwestern University, Evanston, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Mercy Health Riverside, Rockford, Illinois
  - Prairie Heart/St. John's Hospital, Springfield, Illinois
  - Franciscan St. Francis Health, Indianapolis, Indiana
  - Deaconess Heart Group, Newburgh, Indiana
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Kentucky Hospital, Lexington, Kentucky
  - University of Louisville Hospital, Louisville, Kentucky
  - Tulane University Heart and Vascular, New Orleans, Louisiana
  - Ochsner Health System, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - University of Maryland VA, Baltimore, Maryland
  - Johns Hopkins Medical Institution, Baltimore, Maryland
  - White Oak Medical Center, Takoma Park, Maryland
  - St. Elizabeth's Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center (BIDMC), Boston, Massachusetts
  - University of Massachusetts Memorial Hospital, Worcester, Massachusetts
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan
  - University of Michigan Hospital and Health Systems, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Michigan Vascular Center/McLaren- Flint, Flint, Michigan
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Cardiac and Vascular Research Center of Northern Michigan/McLaren Northern Michigan, Petoskey, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Trinity Health/Michigan Heart, Ypsilanti, Michigan
  - Minneapolis Clinic of Neurology, Ltd./North Memorial Medical Center, Golden Valley, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - St. Cloud Hospital, Saint Cloud, Minnesota
  - Cox Medical Center, Springfield, Missouri
  - Mercy Medical Research Institute, Springfield, Missouri
  - John Cochran VA Medical Center, St Louis, Missouri
  - Mercy Hospital, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper University, Camden, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - SUNY Buffalo, Buffalo, New York
  - The Feinstein Institute of Medical Research/Northwell Health, Manhasset, New York
  - Mount Sinai Hospital New York, New York, New York
  - Columbia University Medical Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - St. Francis Hospital, Roslyn, New York
  - Stony Brook University, Stony Brook, New York
  - Crouse Hospital, Syracuse, New York
  - Duke University Medical Center, Durham, North Carolina
  - North Carolina Heart & Vascular Research, Raleigh, North Carolina
  - Coastal Carolina Surgical Associates PA, Wilmington, North Carolina
  - Novant Health/Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Health, Fargo, North Dakota
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Louis Stokes Cleveland VA Medical Center, Cleveland, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Ohio State Medical Center, Columbia, Ohio
  - OhioHealth Research Institute, Columbus, Ohio
  - Jobst Vascular Institute/University of Toledo, Toledo, Ohio
  - Mercy Health St. Vincent Medical Center, Toledo, Ohio
  - St. John Clinical Research Institute, Tulsa, Oklahoma
  - Providence Brain and Spine Institute, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Lehigh Valley Hospital - Network Office of Research, Allentown, Pennsylvania
  - UPMC Altoona, Altoona, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - UPMC Hamot, Erie, Pennsylvania
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - UPMC Presbyterian University Hospital, Pittsburgh, Pennsylvania
  - VA Pittsburgh Healthcare, Pittsburgh, Pennsylvania
  - Pinnacle Health Cardiovascular Institute, Wormleysburg, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Berks Cardiologists / St. Joseph's Medical Center, Wyomissing, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - North Central Heart Institute, Sioux Falls, South Dakota
  - CVA Heart Institute, Kingsport, Tennessee
  - Tennova Healthcare/ Turkey Creek Medical Center, Knoxville, Tennessee
  - Baptist Memorial Hospital, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Seton Medical Center Austin, Austin, Texas
  - Cardiothoracic and Vascular Surgeons, Austin, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Valley Baptist Medical Center, Harlingen, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Utah Hospitals and Clinics, Salt Lake City, Utah
  - George E. Wahlen Department of Veterans Affairs Medical Center, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Inova Fairfax Health Care, Falls Church, Virginia
  - Winchester Medical Center, Winchester, Virginia
  - Overlake Hospital, Bellevue, Washington
  - University of Washington Medicine-Harborview Medical Center, Seattle, Washington
  - VA Puget Sound Health Care System, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
  - Providence Sacred Heart Medical Center, Spokane, Washington
  - West Virginia University, Morgantown, West Virginia
  - Gundersen Clinic, Ltd, La Crosse, Wisconsin
  - University of Wisconsin Hospitals & Clinics, Madison, Wisconsin
- Fiona Stanley Hospital, Perth, Australia
- Canada (5):
  - Vancouver General Hospital, Vancouver, British Columbia
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - St. Michael's Hospital, Toronto, Ontario
  - St. Boniface Hospital, Winnipeg, Ontario
  - CHU de Québec/ Hôpital de l'Enfant-Jésus, Québec, Quebec
- Israel (6):
  - Soroka University Medical Center, Beersheba
  - Soroka University Vascular Surgery, Beersheba
  - Rambam Healthcare, Haifa
  - Hadassah Medical Center, Jerusalem
  - Shaare-Zedek Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
- Hospital Clinic Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brott TG, Howard G, Lal BK, Voeks JH, Turan TN, Roubin GS, Lazar RM, Brown RD Jr, Huston J 3rd, Edwards LJ, Jones M, Clark WM, Chamorro A, Llull L, Mena-Hurtado C, Heck D, Marshall RS, Howard VJ, Moore WS, Barrett KM, Demaerschalk BM, Sangha N, Aronow H, Foster M, Sternbergh WC 3rd, Shawl F, Lanzino G, Rapp J, Tran HS, Ecker R, Mackey A, Ali V, Given C 2nd, Teal P, Kashyap VS, Mukherjee D, Harrigan M, Silverman S, Koopmann M, Wadley VG, Zhang Y, Rhodes JD, Chaturvedi S, Meschia JF; CREST-2 Investigators. Medical Management and Revascularization for Asymptomatic Carotid Stenosis. N Engl J Med. 2026 Jan 15;394(3):219-231. doi: 10.1056/NEJMoa2508800. Epub 2025 Nov 21. PMID 41269206
- [Derived] Meschia JF, Lal B, Roubin G, Turan TN, Howard VJ, Benson RT, Carman K, Howard G, Brott TG. Adapting to Evolving Technologies and Treatment Guidelines in a Procedural Trial: A Qualitative Review of the CREST-2 Experience. Neurology. 2023 May 30;100(22):1060-1066. doi: 10.1212/WNL.0000000000207075. Epub 2023 Feb 6. PMID 36746636
- [Derived] Kamtchum-Tatuene J, Saba L, Heldner MR, Poorthuis MHF, de Borst GJ, Rundek T, Kakkos SK, Chaturvedi S, Topakian R, Polak JF, Jickling GC; Carotid Atherosclerosis and Stroke Collaboration (CASCO). Interleukin-6 Predicts Carotid Plaque Severity, Vulnerability, and Progression. Circ Res. 2022 Jul 8;131(2):e22-e33. doi: 10.1161/CIRCRESAHA.122.320877. Epub 2022 Jun 17. PMID 35713008
- [Derived] Lazar RM, Wadley VG, Myers T, Jones MR, Heck DV, Clark WM, Marshall RS, Howard VJ, Voeks JH, Manly JJ, Moy CS, Chaturvedi S, Meschia JF, Lal BK, Brott TG, Howard G. Baseline Cognitive Impairment in Patients With Asymptomatic Carotid Stenosis in the CREST-2 Trial. Stroke. 2021 Dec;52(12):3855-3863. doi: 10.1161/STROKEAHA.120.032972. Epub 2021 Aug 26. PMID 34433306
- [Derived] Haley W, Shawl F, Charles Sternbergh W 3rd, Turan TN, Barrett K, Voeks J, Brott T, Meschia JF. Non-Adherence to Antihypertensive Guidelines in Patients with Asymptomatic Carotid Stenosis. J Stroke Cerebrovasc Dis. 2021 Aug;30(8):105918. doi: 10.1016/j.jstrokecerebrovasdis.2021.105918. Epub 2021 Jun 18. PMID 34148021
- [Derived] Turan TN, Meschia JF, Chimowitz MI, Roldan A, LeMatty T, Luke S, Breathitt L, Eiland R, Foley J, Brott TG. Mitigating the effects of COVID-19 pandemic on controlling vascular risk factors among participants in a carotid stenosis trial. J Stroke Cerebrovasc Dis. 2020 Dec;29(12):105362. doi: 10.1016/j.jstrokecerebrovasdis.2020.105362. Epub 2020 Sep 30. PMID 33071206
- [Derived] Turan TN, Voeks JH, Chimowitz MI, Roldan A, LeMatty T, Haley W, Lopes-Virella M, Chaturvedi S, Jones M, Heck D, Howard G, Lal BK, Meschia JF, Brott TG. Rationale, Design, and Implementation of Intensive Risk Factor Treatment in the CREST2 Trial. Stroke. 2020 Oct;51(10):2960-2971. doi: 10.1161/STROKEAHA.120.030730. Epub 2020 Sep 21. PMID 32951538
- [Derived] Lal BK, Meschia JF, Roubin GS, Jankowitz B, Heck D, Jovin T, White CJ, Rosenfield K, Katzen B, Dabus G, Gray W, Matsumura J, Hopkins LN, Luke S, Sharma J, Voeks JH, Howard G, Brott TG; CREST-2 Investigators. Factors influencing credentialing of interventionists in the CREST-2 trial. J Vasc Surg. 2020 Mar;71(3):854-861. doi: 10.1016/j.jvs.2019.05.035. Epub 2019 Jul 26. PMID 31353274
- [Derived] Musialek P, Roubin GS. Commentary: Double-Layer Carotid Stents: From the Clinical Need, through a Stent-in-Stent Strategy, to Effective Plaque Isolation... the Journey Toward Safe Carotid Revascularization Using the Endovascular Route. J Endovasc Ther. 2019 Aug;26(4):572-577. doi: 10.1177/1526602819861546. No abstract available. PMID 31303133
- [Derived] Lal BK, Meschia JF, Brott TG. Clinical need, design, and goals for the Carotid Revascularization and Medical Management for Asymptomatic Carotid Stenosis trial. Semin Vasc Surg. 2017 Mar;30(1):2-7. doi: 10.1053/j.semvascsurg.2017.04.004. Epub 2017 Apr 27. PMID 28818255
- [Derived] Demaerschalk BM, Brown RD Jr, Roubin GS, Howard VJ, Cesko E, Barrett KM, Longbottom ME, Voeks JH, Chaturvedi S, Brott TG, Lal BK, Meschia JF, Howard G; CREST-2 Investigators. Factors Associated With Time to Site Activation, Randomization, and Enrollment Performance in a Stroke Prevention Trial. Stroke. 2017 Sep;48(9):2511-2518. doi: 10.1161/STROKEAHA.117.016976. Epub 2017 Aug 2. PMID 28768800
- [Derived] Howard VJ, Meschia JF, Lal BK, Turan TN, Roubin GS, Brown RD Jr, Voeks JH, Barrett KM, Demaerschalk BM, Huston J 3rd, Lazar RM, Moore WS, Wadley VG, Chaturvedi S, Moy CS, Chimowitz M, Howard G, Brott TG; CREST-2 study investigators. Carotid revascularization and medical management for asymptomatic carotid stenosis: Protocol of the CREST-2 clinical trials. Int J Stroke. 2017 Oct;12(7):770-778. doi: 10.1177/1747493017706238. Epub 2017 May 2. PMID 28462683
- See also: CREST-2 Website — http://www.crest2trial.org
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (1):
  • Informed Consent Form (2014-09-24): https://cdn.clinicaltrials.gov/large-docs/17/NCT02089217/ICF_000.pdf